CLINICAL TRIAL: NCT01534221
Title: Randomized Comparison of Outcome of Stenting in Unselected Patients in Everyday Clinical Practice
Brief Title: The COOPerative Establishment for Necessary Investigation in Clinical Outcome After Stenting
Acronym: COPERNICOS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Anders Galloe, Consultant, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COPERNICOS
Record Dates: First submitted 2012-01-30; First posted 2012-02-16 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Ischemic Heart Disease
Keywords: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Study group two (Active Comparator): Endeavor resolute drug eluting stent
  Interventions: Device: Biomatrix drug eluting stent
- Study group three (Active Comparator): The precise selection of brand name depends on negotiations with suppliers and may change during the study period
  Interventions: Device: Biomatrix drug eluting stent
- Study group four (Active Comparator): The precise selection of brand name depends on negotiations with suppliers and may change during the study period
  Interventions: Device: Biomatrix drug eluting stent
- Study group five (Active Comparator): The precise selection of brand name depends on negotiations with suppliers and may change during the study period
  Interventions: Device: Biomatrix drug eluting stent
- Study group one (Active Comparator): The precise selection of brand name depends on negotiations with suppliers and may change during the study period
  Interventions: Device: Biomatrix drug eluting stent

INTERVENTIONS:
Device: Biomatrix drug eluting stent — Biomatrix drug eluting stent
  Other Names: Biomatrix

SUMMARY:
The superiority of a percutaneous coronary intervention (PCI) by one stent over another in terms of clinical outcome is usually documented in large randomized controlled trials (RCT). Although generated from selected study populations these data form the basis for evidence based practice (EBP) in the entire population of patients considered for coronary intervention. An inherent limitation of this approach is that study populations differ significantly from all comers in terms of patient characteristics and prognosis undermining the foundation for extrapolation of trial results to all comers. Furthermore, other trials are based on a "one-fits-all" concept, while the benefits of an "individual-tailored" approach that might be superior, is not investigated.

The Purpose of the current study is to

* Compare clinical outcome between several CE marked drug eluting stents
* Compare clinical outcome between several CE marked bare metal stents
* Compare clinical outcome in all comers with that of the selected study population of RCT's
* Evolve methods to compare clinical outcomes between the generalized "one-fits-all" versus the individualized or "individual-tailored" stent selection approaches

The Method employed is

* All comer PCI registry - single centre
* Randomisation of all eligible patients within the registry to one of several study stent
* Quality assurance in non-randomized population within the registry by periodical alternating the institutional standard stent
* Continuous follow up of all patients included the registry by means of systematic event detection and classification by an independent safety and end point committee
* Assessment of effects on quality of life by heart and health questionnaires

Outcome Measures

Primary endpoints:

* Composite of cardiac death, acute myocardial infraction and target vessel revascularisation
* Stent thrombosis
* A specifically developed Treatment Failure Rate classification

Secondary outcome measures include each of the above, target lesion revascularisation and total death analyzed in a hierarchical fashion at 2, 3, 4 and 5 years.

Tertiary outcome measure is self reported quality of life based on health questionnaires on general health and cardiac symptoms.

Power Calculations An event rate of 20% within 5 years, a relative difference of 25% (an absolute difference of 5%), P< 5%, Power > 80% => 900 patients in each of two treatment arms.

Prespecified Analysis include

1. The MACE rates between stent types
2. The Stent thrombosis rates between stent types
3. The Treatment failure rates between stent types
4. The randomized population versus non-randomized population
5. The individualized versus the generalized Population
6. QOL between stent types

DETAILED DESCRIPTION:
All MACE and stent thromboses are adjudicated by an independent end point and safety committee chaired by Jørgen Jeppesen known from the very same task he executed in the SORT OUT II.

Further question may be answered by the four key investigators:

Steen Carstensen, Anders Galløe, Ole Havndrup, Lars Kjøller-Hansen

ELIGIBILITY:
Inclusion Criteria:

* to enter COPERNICOS registry for quality assessment: Each and every patient assigned to percutaneous coronary intervention will be included.
* to enter COPERNICOS randomization: If the patient fulfil the Helsinki declaration and have a Danish personal security identification number they are asked to give written informed consent to participate in the randomized study arms.

Exclusion Criteria to randomization:

* unconscious patients
* residents in other countries thereby escaping event detection
* patients unable to understand the rationale of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5100 (Estimated)
Dates: Start 2012-03; Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
MACE | Five year
  Major adverse cardiac events defined as a composite of cardiac death, acute myocardial infraction and target vessel revascularisation
Stent thromboses | Five year
  Definite, propable and possible
Treatment failure | Five Years
  A specifically developed Treatment Failure Classification

SECONDARY OUTCOMES:
Death of any cause | One and five years
  Ongoing quality assurance
Self reported health questionnaires on general health and cardiac specific symptoms. | One and five years
Cardiac death | One and five years
Myocardial infarction | One and five years
Target lesion revascularisation | One and five years
Target vessel revascularisation | One and five years
Stent thrombosis | One and five years
Treatment Failure | One and five years

CONTACTS AND LOCATIONS:
Overall Officials: Anders M Galløe, Md.Ph.D., Principal Investigator — Zealand University Hospital; Steen Carstensen, MD, Study Chair — Zealand University Hospital; Ole Havndrup, MD, Study Chair — Zealand University Hospital; Lars Kjøller-Hansen, MD, Study Chair — Zealand University Hospital; Gunnar VH Jensen, MD, Study Director — Zealand University Hospital; Jørgen Jeppesen, MD, Study Director — Glostrup University Hospital, Copenhagen
Locations (1):
- Roskilde County Hospital, Roskilde, Denmark